CLINICAL TRIAL: NCT04365088
Title: Evaluation of the Effects of Pre-operative Deflazacort on Post-operative Pain, Edema and Trismus in Impacted Lower Third Molar Surgery
Brief Title: Evaluation of the Effects of Pre-operative Deflazacort on Post-operative Pain, Edema and Trismus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, levent Cigerim, Head of Oral and Maxillofacial Surgery Department, Yuzuncu Yil University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19.07.2017/06
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Impacted Third Molar Tooth
Keywords: deflazacort; pain; edema; trismus
MeSH Terms: conditions — Pain; Edema; Trismus | interventions — deflazacort; Tablets; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deflazacort (Experimental): Deflazacort is a glucocorticoid used as an anti-inflammatory drug. We used deflazacort 30 mg tablet. Patient took a pill once preoperatively (1 hour ago) in third molar surgery.
  Interventions: Drug: Deflazacort 30 MG Oral Tablet
- Sugar pill (Placebo Comparator): Placebo is an inert substance or treatment which is designed to have no therapeutic value. Patients took sugar pill for plasebo once one hour before operation.
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Deflazacort 30 MG Oral Tablet — After the taken a deflazacort pill once preoperatively (one hour ago), local anesthesia was obtained using 2 ml articaine hydrochloride 40 mg/ml with epinephrine 0.01 mg/ml . The horizontal incision was made with no. 15 scalpel blade and a full thickness mucoperiosteal flap was raised. In all surgical procedures, bone removal and/or tooth sectioning were performed under sterile saline irrigation. Following the extraction, granulation tissues were removed, and bleeding was controlled. Finally, the mucoperiosteal flap was repositioned by 3.0 silk sutures.
  Other Names: FLANTADIN 30 MG 10 TABLET
  Arms: Deflazacort
Drug: Sugar pill — Sugar pill
  Arms: Sugar pill

SUMMARY:
Removal of impacted lower third molar teeth is one of the most common oral surgical procedures, and these operations often lead to various complications in patients. Antibiotics, analgesics and/or anti-inflammatory drugs are prescribed for the treatment of complications encountered. Anti-inflammatory is the property of a substance or treatment that reduces inflammation or swelling. Anti-inflammatory drugs make up about half of analgesics, remedying pain by reducing inflammation as opposed to opioids, which affect the central nervous system to block pain signaling to the brain. Based on this information, in this study, it is aimed to evaluate the effects of deflazacort preoperatively on the postoperative pain, swelling and trismus.

ELIGIBILITY:
Inclusion Criteria:

* absence of any systemic disease,
* having bilateral impacted mandibular third molar teeth in a similar position
* absence of allergy to any of the drugs used in the study,
* absence of pregnancy/lactating state,
* no history of any medication use during at least 2 week before the operation.

Exclusion Criteria:

* not regularly coming to the controls,
* not using their medicines regularly,
* using any additional medication that may affect the outcome of the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain | Postoperative 1st day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 2nd day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Edema | Postoperative 2nd day
  Postoperative edema was evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion) which was measured with using thread and millimeter ruler.
Postoperative Trismus | Postoperative 2nd day
  Postoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.
Postoperative Pain | Postoperative 3d day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 4th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 5th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 6th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Pain | Postoperative 7th day
  Patients were requested to mark their pain intensity on a pain assessment form using a visual analoge scale (VAS) ranging between 0 (no pain) to 10 (most severe pain).
Postoperative Edema | Postoperative 7th day
  Postoperative edema was evaluated by the distance between predetermined facial anatomic landmarks (from the mandibular angle to lateral corner of the eye, base of the nose, labial commissura, and soft tissue pogonion) which was measured with using thread and millimeter ruler.
Postoperative Trismus | Postoperative 7th day
  Postoperative trismus was evaluated by the maximum distance between the incisive borders of the upper and lower right incisive teeth which was measured with a caliper.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Tuşba, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No